CLINICAL TRIAL: NCT01408342
Title: Low-doses Alemtuzumab and Rituximab Combination as First Line Treatment in Aplastic Anemia
Brief Title: Alemtuzumab and Rituximab in Aplastic Anemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE11015; AA
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Aplastic Anemia
Keywords: Alemtuzumab; Rituximab; Aplastic anemia; cyclosporine
MeSH Terms: conditions — Anemia, Aplastic | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab, Alemtuzumab (Other)
  Interventions: Drug: Alemtuzumab and Rituximab

INTERVENTIONS:
Drug: Alemtuzumab and Rituximab — * Alemtuzumab 10 mg (5 mg/m2 in patients under 30 kg weight) subcutaneous days 1,2 and 3
  * Rituximab 100 mg (50 mg/m2 in patients under 30 kg weight)intravenous days 4,11,18,25
  * Cyclosporine 3 mg/kg starting day 21
  Other Names: Kikuzubam; Mabthera; Mabcampath; Campath

SUMMARY:
The purpose of the study is to evaluate the efficacy of combination of alemtuzumab and rituximab as first line therapy in aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aplastic anemia diagnosis

Exclusion Criteria:

* Patients with prior treatment with monoclonal antibodies and/or antithymocyte globulin.
* Patients with a diagnosis or history of HIV/AIDS, Hepatitis B, Hepatitis C, Cytomegalovirus.
* Patients who do not agree to sign a Letter of Informed Consent.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of alemtuzumab and rituximab in aplastic anemia. | 12 months
  Evaluate the hematological response after the administration of alemtuzumab and rituximab

SECONDARY OUTCOMES:
Measuring the side effects of alemtuzumab and rituximab combination through clinical evaluation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez Almaguer, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hospital Universitario, Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Young NS, Maciejewski J. The pathophysiology of acquired aplastic anemia. N Engl J Med. 1997 May 8;336(19):1365-72. doi: 10.1056/NEJM199705083361906. No abstract available. PMID 9134878
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Gomez-Almaguer D, Jaime-Perez JC, Garza-Rodriguez V, Chapa-Rodriguez A, Tarin-Arzaga L, Herrera-Garza JL, Ruiz-Arguelles GJ, Lopez-Otero A, Gonzalez-Llano O, Rodriguez-Romo L. Subcutaneous alemtuzumab plus cyclosporine for the treatment of aplastic anemia. Ann Hematol. 2010 Mar;89(3):299-303. doi: 10.1007/s00277-009-0816-5. Epub 2009 Aug 25. PMID 19705116
- [Background] Takamatsu H, Yagasaki H, Takahashi Y, Hama A, Saikawa Y, Yachie A, Koizumi S, Kojima S, Nakao S. Aplastic anemia successfully treated with rituximab: the possible role of aplastic anemia-associated autoantibodies as a marker for response. Eur J Haematol. 2011 Jun;86(6):541-5. doi: 10.1111/j.1600-0609.2011.01612.x. PMID 21418330
- [Background] Gomez-Almaguer D, Solano-Genesta M, Tarin-Arzaga L, Herrera-Garza JL, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Jaime-Perez JC. Low-dose rituximab and alemtuzumab combination therapy for patients with steroid-refractory autoimmune cytopenias. Blood. 2010 Dec 2;116(23):4783-5. doi: 10.1182/blood-2010-06-291831. Epub 2010 Sep 14. PMID 20841509
- [Background] Risitano AM, Selleri C, Serio B, Torelli GF, Kulagin A, Maury S, Halter J, Gupta V, Bacigalupo A, Socie G, Tichelli A, Schrezenmeier H, Marsh J, Passweg J, Rotoli B; Working Party Severe Aplastic Anaemia (WPSAA) of the European Group for Blood and Marrow Transplantation (EBMT). Alemtuzumab is safe and effective as immunosuppressive treatment for aplastic anaemia and single-lineage marrow failure: a pilot study and a survey from the EBMT WPSAA. Br J Haematol. 2010 Mar;148(5):791-6. doi: 10.1111/j.1365-2141.2009.08027.x. Epub 2009 Dec 7. PMID 19995389